CLINICAL TRIAL: NCT05193331
Title: 3% Diquafosol Topical Ophthalmic Solution in Diabetic Patients With Dry Eye
Brief Title: Use of 3% Diquafosol Topical Ophthalmic Solution for Diabetic Dry Eye
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: He Eye Hospital (Other)
Collaborators: Santen Pharmaceutical(China) Co.,LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P-DBDED-DQS-2021
Record Dates: First submitted 2022-01-02; First posted 2022-01-14 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Diabetic Eye Problems
Keywords: Dry eye; Diquafosol; Hyaluronate; Diabetic dry eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Prospective study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DQS group (Experimental): Participants in DQS group will be administered one drop of 3% DQS (Diquas, Santen Pharmaceutical Co., Ltd., Osaka, Japan) six times per day for 4 weeks (28 days).
  Interventions: Drug: 3% Diquafosol tetrasodium

INTERVENTIONS:
Drug: 3% Diquafosol tetrasodium — 3% Diquafosol tetrasodium eye drops will be used to assess its usefulness in diabetic dry eye symptoms
  Other Names: Diquas

SUMMARY:
Diquafosol ophthalmic solution (DQS) stimulates P2Y2 receptors on the ocular surface, which enhances mucin secretion from goblet cells. Therefore, tear film stability and hydration of the ocular surface can be achieved independent from lacrimal glands function. This prospective, open label pilot study will include 140 eyes of 70 diabetic patients diagnosed with DED and will be consecutively assigned to DQS (n=140 eyes). Participants in the DQS group will receive 3% Diquafosol ophthalmic solution. The dosage of 3% Diquafosol will be one drop, six times per day for 4 weeks. Tear film lipid layer (TFLL), non-invasive breakup time (NITBUT), corneoconjunctival staining score (CS), meibum gland (MG), conjunctival hyperemia (RS score), ocular surface disease index (OSDI) will be assessed and compared at baseline, day-14, and day-28.

DETAILED DESCRIPTION:
This study will be conducted in compliance with the tenets of the Declaration of Helsinki and the Institutional Review Board of He Eye Specialist Hospital, Shenyang, China [ethics approval number: IRB(2022)K002.01]

Type 2 diabetes mellitus (T2DM) is a prevalent chronic metabolic illness that causes relative insulin insufficiency in target organs owing to pancreatic β-cell dysfunction and insulin resistance. Shift to sedentary lifestyle, ageing population and obesity has significantly contributed to the global rise in the prevalence of T2DM. In 2019 the prevalence of diabetes was documented to be 9.3% (463 million people) and in 2030 it is estimated to rise to 10.2% (578 million) and T2DM accounts for approximately 90% of all diabetic occurrence. Negative alterations to the tear film, corneal epithelium, corneal endothelium, and corneal nerves have been observed in 47-64% of patients with diabetes. Ocular surface manifestation of signs and symptoms secondary to DM has been termed as diabetic keratopathy (DK). DK has been documented to increase central corneal thickness[6], decrease in endothelial cell density, leads of superficial punctate keratitis[8], delay and impede wound repair[9], and decrease in corneal sensitivity due to neuropathy. Additionally, DM patients have also been noted to have compromised tear quantity and quality due to conjunctival goblet cell loss as documented on cytologic analysis. Goblet cells secrete mucin, which stabilizes the tear film, minimizes tear evaporation, and reduces mechanical friction. Goblet cell loss in animal models suggests that it disrupts the ocular surface's immune tolerance and increased expression of inflammatory cytokines in the conjunctiva. 0.1% hyaluronate (HA) used in artificial tears have been reported to promote corneal re-epithelium and improve corneal healing.

Diquafosol tetrasodium is a dinucleotide polyphosphate which a purinoceptor agonist, when administered to the ocular surface, it binds to P2Y2 receptors and stimulates mucin and tear secretion. The corneal epithelium, conjunctival epithelium, lacrimal gland ductal epithelium, meibomian gland sebaceous cells, and meibomian gland ductal cells all express the P2Y2 receptor. Subsequently, enhanced secretion of mucin and tear secretion due to Diquafosol tetrasodium ophthalmic solution (DQS) stabilize the tear film, minimizes tear evaporation, and reduces mechanical friction thereby protecting the corneal epithelium [23]. Various reports have concluded that that 3% DQS is effective in the treatment of dry eye disease and the year 2020's findings suggest that DQS improves corneal epithelial damage in T2DM rat model.

However, the effect of DQS on the tear film of T2DM humans has not been previously assessed. Therefore, the purpose s to assess subjective and objective diabetic dry eye findings after using 3% DQS topical eye drops.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinical diagnosed and confirmed with type 2 diabetes for one year or more
* Able and willing to comply with the treatment/follow-up schedule
* Bilateral signs and symptoms of dry eye disease

Exclusion Criteria:

* Participants with systemic immune-mediated illnesses, such as secondary Sjögren's syndrome or graft-versus-host disease
* Patients using topical medication(s) for the treatment of ocular disorders such as glaucoma or allergic conjunctivitis were excluded from the study.
* Previous ocular surgery or trauma
* 1-month history of blepharal and periorbital skin disease or allergies
* Severe dry eyes with corneal epithelial defect
* Limbic keratitis
* Pterygium
* Corneal neovascularization
* Glaucoma
* Breastfeeding
* Rheumatic immune systemic diseases
* Herpes zoster infection
* Pregnant women
* Allergic to fluorescein
* Contact lens wearers

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Non-invasive tear break-up time | Day-0 (baseline), 4-weeks and 8-weeks
  Non-invasive initial tear film breaking time will be assessed using the Keratograph 5M (Oculus, Germany) topographer. Three sequentially readings will be captured, and the median value will be included in the final analysis. The median value will be recorded.

SECONDARY OUTCOMES:
Fluorescein and lissamine conjunctival and cornea staining | Day-0 (baseline), 4-weeks and 8-weeks
  Fluorescein and lissamine staining of the ocular surface will be divided into three zones comprising nasal conjunctival, corneal, and temporal conjunctival areas. The staining score ranged from 0 to 3 for each zone, yielding a total score of 0-9 for the ocular surface (Uchino et al., 2012).
Tear Film Lipid Layer Score | Day-0 (baseline), 4-weeks and 8-weeks
  Tear Film Lipid Layer interferometry will be assessed using DR-1 (Kowa, Nagoya, Japan).
  - Tear Film Lipid Layer will be scored as follows: grade 1, somewhat gray color, uniform distribution; grade 2, somewhat gray color, nonuniform distribution; grade 3, a few colors, nonuniform distribution; grade 4, many colors, nonuniform distribution; grade 5, corneal surface partially exposed.
Corneal Sensitivity Score | Day-0 (baseline), 4-weeks and 8-weeks
  Corneal Sensitivity Score measured with Cochet-Bonnet esthesiometer (in mm filament length) two times (the measurements will be done immediately before starting the medication, including 3 measurements each time.
MMP-9 detection | Day-0 (baseline), 4-weeks and 8-weeks
  InflammaDry, (Rapid Pathogen Screening Inc., Sarasota, FL, USA) is a patented and proprietary modification of a traditional lateral flow device and uses direct sampling microfiltration technology. Two antigen-specific antibodies capture MMP-9 antigens in the sample, and this complex is captured in a proprietary mode at the test result line, giving rise to a visually observable signal.
Tear meniscus height | Day-0 (baseline), 4-weeks and 8-weeks
  Non-invasive first tear film breakup time using the Keratograph 5M (Oculus, Germany) topographer will be measured three times consecutively and the median value was recorded. of the three values was calculated.
Conjunctival hyperemia (RS score) | Day-0 (baseline), 4-weeks and 8-weeks
  Conjunctival hyperemia (RS score) will be assessed by keratograph image (Oculus, Germany) of 1156*873 pixels, redness score (RS) (accurate to 0.1 U) was displayed on the computer screen that ranged from 0.0 to 4.0.
Meibomian gland function and secretion quality | Day-0 (baseline), 4-weeks and 8-weeks
  Meibum quality will be assessed under a slit-lamp:
  Five meibomian gland in the middle parts of the eyelid will be assessed using a scale of 0 to 3 for each gland (0 represented clear meibum; 1 represented cloudy meibum; 2 represented cloudy and granular meibum; and 3 represented thick, toothpaste like consistency meibum).
Corneal nerves and immune/inflammatory cells change | Day-0 (baseline), 4-weeks and 8-weeks
  HRT III RCM, (Heidelberg Engineering GmbH, Dossenheim, Germany) will be used to record corneal nerves and immune/inflammatory cells change. A total of 5-8 sequence/volume scans were taken from the center of each cornea, focusing on all corneal layers: superficial, intermediate, and basal epithelial layers, sub-basal nerve plexus, anterior, central and posterior stroma, and endothelium. Special attention was given to the basal epithelial layer and sub-basal nerve plexus area to evaluate the nerve plexi and epithelial DC density. Three representative images of the sub-basal nerve plexus and epithelial DCs were selected for analysis for each eye, considering criteria such as whole image in the same layer, best focus and good contrast.
Dry eye Questionnaire Score | Day-0 (baseline), 4-weeks and 8-weeks
  Chinese translated version of the questionnaire will be used to assess the subjective dry eye symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel E Pazo, PhD, Study Chair — He Eye Hospital, Shenyang, China
Locations (1):
- He Eye Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chatterjee S, Khunti K, Davies MJ. Type 2 diabetes. Lancet. 2017 Jun 3;389(10085):2239-2251. doi: 10.1016/S0140-6736(17)30058-2. Epub 2017 Feb 10. PMID 28190580
- [Result] Weisman A, Fazli GS, Johns A, Booth GL. Evolving Trends in the Epidemiology, Risk Factors, and Prevention of Type 2 Diabetes: A Review. Can J Cardiol. 2018 May;34(5):552-564. doi: 10.1016/j.cjca.2018.03.002. Epub 2018 Mar 13. PMID 29731019
- [Result] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Result] Abdelkader H, Patel DV, McGhee CNj, Alany RG. New therapeutic approaches in the treatment of diabetic keratopathy: a review. Clin Exp Ophthalmol. 2011 Apr;39(3):259-70. doi: 10.1111/j.1442-9071.2010.02435.x. Epub 2011 Apr 4. PMID 20973888
- [Result] Vieira-Potter VJ, Karamichos D, Lee DJ. Ocular Complications of Diabetes and Therapeutic Approaches. Biomed Res Int. 2016;2016:3801570. doi: 10.1155/2016/3801570. Epub 2016 Mar 28. PMID 27119078
- [Result] El-Agamy A, Alsubaie S. Corneal endothelium and central corneal thickness changes in type 2 diabetes mellitus. Clin Ophthalmol. 2017 Mar 2;11:481-486. doi: 10.2147/OPTH.S126217. eCollection 2017. PMID 28280298
- [Result] Lee JS, Oum BS, Choi HY, Lee JE, Cho BM. Differences in corneal thickness and corneal endothelium related to duration in diabetes. Eye (Lond). 2006 Mar;20(3):315-8. doi: 10.1038/sj.eye.6701868. PMID 15832184
- [Result] Inoue K, Okugawa K, Amano S, Oshika T, Takamura E, Egami F, Umizu G, Aikawa K, Kato S. Blinking and superficial punctate keratopathy in patients with diabetes mellitus. Eye (Lond). 2005 Apr;19(4):418-21. doi: 10.1038/sj.eye.6701497. PMID 15286669
- [Result] Shih KC, Lam KS, Tong L. A systematic review on the impact of diabetes mellitus on the ocular surface. Nutr Diabetes. 2017 Mar 20;7(3):e251. doi: 10.1038/nutd.2017.4. PMID 28319106
- [Result] Murphy PJ, Patel S, Kong N, Ryder RE, Marshall J. Noninvasive assessment of corneal sensitivity in young and elderly diabetic and nondiabetic subjects. Invest Ophthalmol Vis Sci. 2004 Jun;45(6):1737-42. doi: 10.1167/iovs.03-0689. PMID 15161834
- [Result] Dogru M, Katakami C, Inoue M. Tear function and ocular surface changes in noninsulin-dependent diabetes mellitus. Ophthalmology. 2001 Mar;108(3):586-92. doi: 10.1016/s0161-6420(00)00599-6. PMID 11237914
- [Result] Sagdik HM, Ugurbas SH, Can M, Tetikoglu M, Ugurbas E, Ugurbas SC, Alpay A, Ucar F. Tear film osmolarity in patients with diabetes mellitus. Ophthalmic Res. 2013;50(1):1-5. doi: 10.1159/000345770. Epub 2013 Feb 22. PMID 23445780
- [Result] Barbosa FL, Xiao Y, Bian F, Coursey TG, Ko BY, Clevers H, de Paiva CS, Pflugfelder SC. Goblet Cells Contribute to Ocular Surface Immune Tolerance-Implications for Dry Eye Disease. Int J Mol Sci. 2017 May 5;18(5):978. doi: 10.3390/ijms18050978. PMID 28475124
- [Result] Marko CK, Menon BB, Chen G, Whitsett JA, Clevers H, Gipson IK. Spdef null mice lack conjunctival goblet cells and provide a model of dry eye. Am J Pathol. 2013 Jul;183(1):35-48. doi: 10.1016/j.ajpath.2013.03.017. Epub 2013 May 10. PMID 23665202
- [Result] Park Y, Song JS, Choi CY, Yoon KC, Lee HK, Kim HS. A Randomized Multicenter Study Comparing 0.1%, 0.15%, and 0.3% Sodium Hyaluronate with 0.05% Cyclosporine in the Treatment of Dry Eye. J Ocul Pharmacol Ther. 2017 Mar;33(2):66-72. doi: 10.1089/jop.2016.0086. Epub 2016 Dec 8. PMID 27929721
- [Result] Jeon HS, Hyon JY. The Efficacy of Diquafosol Ophthalmic Solution in Non-Sjogren and Sjogren Syndrome Dry Eye Patients Unresponsive to Artificial Tear. J Ocul Pharmacol Ther. 2016 Sep;32(7):463-8. doi: 10.1089/jop.2015.0081. Epub 2016 Jun 13. PMID 27294831
- [Result] Jumblatt JE, Jumblatt MM. Regulation of ocular mucin secretion by P2Y2 nucleotide receptors in rabbit and human conjunctiva. Exp Eye Res. 1998 Sep;67(3):341-6. doi: 10.1006/exer.1998.0520. PMID 9778415
- [Result] Dota A, Sakamoto A, Nagano T, Murakami T, Matsugi T. Effect of Diquafosol Ophthalmic Solution on Airflow-Induced Ocular Surface Disorder in Diabetic Rats. Clin Ophthalmol. 2020 Apr 1;14:1019-1024. doi: 10.2147/OPTH.S242764. eCollection 2020. PMID 32280196
- [Result] Kulkarni AA, Trousdale MD, Stevenson D, Gukasyan HJ, Shiue MH, Kim KJ, Read RW, Lee VH. Nucleotide-induced restoration of conjunctival chloride and fluid secretion in adenovirus type 5-infected pigmented rabbit eyes. J Pharmacol Exp Ther. 2003 Jun;305(3):1206-11. doi: 10.1124/jpet.103.049221. Epub 2003 Mar 20. PMID 12649304
- [Result] Cowlen MS, Zhang VZ, Warnock L, Moyer CF, Peterson WM, Yerxa BR. Localization of ocular P2Y2 receptor gene expression by in situ hybridization. Exp Eye Res. 2003 Jul;77(1):77-84. doi: 10.1016/s0014-4835(03)00068-x. PMID 12823990
- [Result] Tanioka H, Kuriki Y, Sakamoto A, Katsuta O, Kawazu K, Nakamura M. Expression of the P2Y(2) receptor on the rat ocular surface during a 1-year rearing period. Jpn J Ophthalmol. 2014 Nov;58(6):515-21. doi: 10.1007/s10384-014-0342-4. Epub 2014 Sep 2. PMID 25179431
- [Result] Yuko, T.S.; NAKAMURA, M. Stimulatory Effect of Diquafosol Tetrasodium on the Expression of Membrane-Binding Mucin Genes in Cultured Human Corneal Epithelial Cells. Journal of the eye 2011, 28, 425-429.
- [Result] Kaido M, Kawashima M, Shigeno Y, Yamada Y, Tsubota K. Randomized Controlled Study to Investigate the Effect of Topical Diquafosol Tetrasodium on Corneal Sensitivity in Short Tear Break-Up Time Dry Eye. Adv Ther. 2018 May;35(5):697-706. doi: 10.1007/s12325-018-0685-1. Epub 2018 Apr 18. PMID 29671255
- [Result] Ji YW, Kim HM, Ryu SY, Oh JW, Yeo A, Choi CY, Kim MJ, Song JS, Kim HS, Seo KY, Kim KP, Lee HK. Changes in Human Tear Proteome Following Topical Treatment of Dry Eye Disease: Cyclosporine A Versus Diquafosol Tetrasodium. Invest Ophthalmol Vis Sci. 2019 Dec 2;60(15):5035-5044. doi: 10.1167/iovs.19-27872. PMID 31800960
- [Result] Amano S, Inoue K. Effect of topical 3% diquafosol sodium on eyes with dry eye disease and meibomian gland dysfunction. Clin Ophthalmol. 2017 Sep 14;11:1677-1682. doi: 10.2147/OPTH.S148167. eCollection 2017. PMID 29075094
- [Result] Ohashi Y, Munesue M, Shimazaki J, Takamura E, Yokoi N, Watanabe H, Nomura A, Shimada F. Long-Term Safety and Effectiveness of Diquafosol for the Treatment of Dry Eye in a Real-World Setting: A Prospective Observational Study. Adv Ther. 2020 Feb;37(2):707-717. doi: 10.1007/s12325-019-01188-x. Epub 2019 Dec 13. PMID 31834617
- [Derived] Qin G, Chen J, Li L, Qi Y, Chen Y, Zhang Q, Wu Y, You Y, Yang L, Guo N, Moutari S, Bu S, Moore JE, Xu L, He W, Yu S, He X, Pazo EE. Effects of Diquafosol Sodium Ophthalmic Solution on Tear Film Matrix Metallopeptidase-9 and Corneal Nerve Density in Patients with Type 2 Diabetic Dry Eye. J Ocul Pharmacol Ther. 2024 Jul-Aug;40(6):370-378. doi: 10.1089/jop.2023.0098. Epub 2023 Dec 13. PMID 38100078
- [Derived] Qin G, Chen J, Li L, Qi Y, Zhang Q, Wu Y, You Y, Yang L, Moore J, Xu L, He W, Yu S, Pazo EE, He X. Relationship between ocular surface pain and corneal nerve loss in dry eye diabetics: a cross-sectional study in Shenyang, China. BMJ Open. 2023 Sep 26;13(9):e076932. doi: 10.1136/bmjopen-2023-076932. PMID 37751961